CLINICAL TRIAL: NCT06523660
Title: A Randomized, Control Trial of Executive Function Training for Korean Kindergartners With Autism Spectrum Disorder
Brief Title: Improving Executive Function in Korean Children With Autism
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, So Hyun Kim, Associate Professor, Korea University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-2024-0026; 00209635 (Other Grant/Funding Number: National Research Foundation of Korea)
Record Dates: First submitted 2024-07-17; First posted 2024-07-26 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Children will receive the EF training intervention, which will be delivered in a telehealth format across 10 sessions (1 1-hour session per week for 10 weeks), targeting core EF components including inhibitory control, attention shifting, and working memory. Accompanied parent coaching will be provided to enhance children's generalization of EF skill attainment.
  Interventions: Behavioral: CHUCK CHUCK SKILLS: CHild's Understanding of Cognitive sKills
- Control Group (Active Comparator): Group-based parent psychoeducation will be provided to the control group. This program will also be delivered in a telehealth format across 10 sessions (1 1-hour session per week for 10 weeks) and will cover a broad range of information relevant to ASD.
  Interventions: Behavioral: Parent Psychoeducation

INTERVENTIONS:
Behavioral: CHUCK CHUCK SKILLS: CHild's Understanding of Cognitive sKills — The intervention will consist of an online EF training that will be delivered across 10 sessions (one 1 hour session per week for ten weeks). It will target core EF components including inhibitory control, attention shifting, and working memory in children with Autism Spectrum Disorder aged 5 to 7 years. It will also provide strategies (e.g., behavioral principles, compliance training) for promoting behavioral regulation and emotion regulation in these children. Accompanied parent coaching will be provided to enhance children's generalization of EF skill attainment.
  Arms: Intervention Group
Behavioral: Parent Psychoeducation — Group-based parent psychoeducation, which consists of 10 sessions, 1-hour weekly program delivered via telehealth, will be provided to the control group.
  Arms: Control Group

SUMMARY:
The purpose of this randomized controlled study is to evaluate the acceptability, feasibility, and preliminary efficacy of an executive function (EF) training intervention for 5- to 7-year-old autistic children in South Korea. This study will have three aims: (1) to assess the acceptability and feasibility of the EF intervention with children with ASD; (2) to examine clinically important effects of the intervention using multimodal methods combining lab-based behavioral tasks and novel electrophysiological measures; and (3) to determine whether the effects are generalized to everyday EF skills in real-world settings using parent-ratings.

DETAILED DESCRIPTION:
The ability to self-monitor and flexibly adapt behavior in response to internal or external changes refers to neurocognitive processes known as executive function (EF). EF impairments, such as inflexible problem-solving, attention-shifting difficulties, and challenges in goal-directed behavior planning, are consistently identified as core cognitive deficits in autism spectrum disorder (ASD). Early life EF deficits can lead to negative social and academic outcomes, including poor school performance, externalizing behaviors, antisocial conduct, and adverse adult outcomes. Therefore, EF has become a significant focus for interventions, yet few studies have investigated EF interventions in ASD. Evidence-based interventions targeting EF are critically needed.

The purpose of this randomized controlled study is to evaluate the effectiveness of an online EF training intervention for 5- to 7-year-old children with ASD in South Korea, where intervention services, especially during school transition periods, are extremely limited. The project has three scientific goals: (1) assess the acceptability and feasibility of the EF intervention for children with ASD; (2) examine the clinically important effects of the intervention using multimodal methods combining lab-based behavioral tasks and novel electrophysiological measures; and (3) determine whether the effects generalize to everyday EF skills in real-world settings using parent-ratings.

The investigators will recruit 40 Korean children with ASD during school transition (20 randomly assigned to the intervention, 20 to the control). Children in the intervention group will participate in a 10-week online training program and will be administered outcome measures, including physiological measures, lab-based behavior, and parent-reports of clinical functioning, at three time points (i.e., pre-intervention, 1-week after the completion of the intervention, and 3-months after the completion of the intervention). Parent coaching will be provided to enhance the generalization of EF skills. The control group will receive group-based parent psychoeducation. This work has the potential to significantly improve EF skills and functional outcomes for autistic children, addressing the urgent need for targeted interventions for the underserved population in South Korea.

ELIGIBILITY:
Inclusion Criteria:

* Previous medical diagnosis of ASD, confirmed by Autism Diagnostic Observation Schedule, Second Edition (ADOS-2)
* Non-verbal IQ (NVIQ) equal to or above 85
* Verbal children (with flexible phrases or complex sentences)

Exclusion Criteria:

* NVIQ below 85
* Presence of medical disorders or injuries with implications for the central nervous system or that require medications that alter EEG processes such as anticonvulsants
* Presence of significant sensory or motor impairment
* Presence of major physical anomalies

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Executive Function (EF) Touch | pre-intervention, post-intervention (1 week after the completion of the intervention), 3-month follow-up (3 months after the completion of the intervention)
  Executive Function (EF) Touch is a child-friendly computerized assessment of executive function skills, administered on a touch-screen tablet. The use of Executive Function Touch will allow the investigators to target fine-grained, multiple EF domains, including inhibitory control ("Spatial Conflict Arrows"), working memory ("Pick the Picture"), and attention shifting ("Something's the Same). The investigators will use a proportion of correct trials from each task as the outcome measure, with higher scores indicating a better performance on the task (minimum = 0, maximum = 1).
Head-Toes-Knees-Shoulders (HTKS) | pre-intervention, post-intervention (1 week after the completion of the intervention), 3-month follow-up (3 months after the completion of the intervention)
  Head-Toes-Knees-Shoulders (HTKS) is a behavioral task that measures self-regulation in children and consists of short tasks suitable for children 4-8 years of age, with higher scores indicating a better performance (minimum = 0, maximum = 118).
Stroop Color and Word Test Children's Version (Stroop) | pre-intervention, post-intervention (1 week after the completion of the intervention), 3-month follow-up (3 months after the completion of the intervention)
  The Stroop test is a neuropsychological measure for assessing the efficiency of inhibitory control. Participants are asked to read 1) the Word page where names of colors are printed in black 2) the Color page where patches labeled as 'XXXX' are printed in different colors 3) the Color-Word page where names of colors are printed in inconsistent colors (ex. the word "red" is printed in blue, and participants need to read out the color "blue" instead of the word "red".). The number of items correctly read within 45 seconds for each page is recorded.
Korean-Boston Naming Test-Children's Version (K-BNT-C) | pre-intervention, post-intervention (1 week after the completion of the intervention), 3-month follow-up (3 months after the completion of the intervention)
  The Korean-Boston Naming Test-Children's Version assesses not only the "word processing", but also the "visuospatial perception" of the pictures. Participants are shown black-and-white pictures of objects and asked to name them.
Children's Color Trail Making Test (CCTT) | pre-intervention, post-intervention (1 week after the completion of the intervention), 3-month follow-up (3 months after the completion of the intervention)
  Children's Color Trail Making Test (CCTT) consists of two subscales: CCTT-1, which requires perceptual tracking, sustained attention, and fine motor skills, and CCTT-2, which requires divided attention, sequential processing, and inhibition/disinhibition in addition to the first three skills. Participants are asked to connect circles with numbers and colors in order, and the time spent to complete each task is recorded.
The Behavior Rating Inventory of Executive Function (BRIEF) | pre-intervention, post-intervention (1 week after the completion of the intervention), 3-month follow-up (3 months after the completion of the intervention)
  The BRIEF is a standardized parent report measure where parents rate the frequency of their child's EF challenges within everyday contexts, such as home and other community settings. The BRIEF results in scores that reflect the child's level of EF dysfunction, with higher scores indicating more EF challenges. The BRIEF consists of 63 items, with each item rated on a 3-point Likert scale (1 = Never, 2 = Sometimes, 3 = Often). In this study, the investigators will use T-scores from clinical scales (e.g., Inhibit, Shift, Working Memory) of the BRIEF (M=50, SD=10), as well as Global Executive Composite, an overall summary score that incorporates all the clinical scales of the BRIEF.
Emotion Dysregulation Inventory (EDI) | pre-intervention, post-intervention (1 week after the completion of the intervention), 3-month follow-up (3 months after the completion of the intervention)
  The Emotion Dysregulation Inventory (EDI) is a parent-report questionnaire that assesses emotion regulation difficulties of children, rated on a five-point scale from "not at all" to "very severe." The EDI results in scores that reflect the child's level of emotion regulation dysfunction, with higher scores representing more emotion regulation challenges. The investigators will use a 30-item full version of the EDI, which consists of 24 items related to Reactivity and 6 items related to Dysphoria. Raw scores of the Reactivity scale range from 0 to 96. Raw scores of the Dysphoria range from 0 to 24.
EF Training Program Feasibility Survey | post-intervention (1 week after the completion of the intervention)
  This will be completed by the parents at the end of the intervention program to assess whether the intervention was feasible for the participants. It will include items related to practicality of the program such as 'zoom was easy to operate' and 'I was able to find time to do homework with my child', and parents will provide answers on a likert scale.
EF Training Program Acceptability Survey | post-intervention (1 week after the completion of the intervention)
  This will be completed by the parents at the end of the intervention program to assess whether the intervention was acceptable and satisfying to the participants. It will include items such as 'I benefit from intervention sessions with the interventionist' and parents will provide answers on a likert scale.

SECONDARY OUTCOMES:
Vineland Adaptive Behavior Scale (VABS) | pre-intervention, post-intervention (1 week after the completion of the intervention), 3-month follow-up (3 months after the completion of the intervention)
  The VABS is a standardized parent report to measure children's social skills, communication, and adaptive behavior. Higher scores on each subscale indicate better adaptive function.
Penn Interactive Peer Play Scale (PIPPS) | pre-intervention, post-intervention (1 week after the completion of the intervention), 3-month follow-up (3 months after the completion of the intervention)
  The PIPPS is a play behavior assessment developed to understand children's interactions with peers. It consists of three subscales: play interaction, play disruption, play disconnection. 1) Play Interaction is an indication of children's play strengths and includes such behaviors as comforting and helping other children, showing creativity in play, and encouraging others to join play. 2) Play Disruption describes aggressive, antisocial behaviors that interfere with on-going peer play interactions. 3) Play Disconnection reflects withdrawn behavior and non-participation in peer play.
Children's Behavior Checklist (CBCL) | pre-intervention, post-intervention (1 week after the completion of the intervention), 3-month follow-up (3 months after the completion of the intervention)
  The CBCL is a standardized behavior rating scale informed by parents and / or teachers for assessing child behavior. It is scored on a three-point Likert scale (0=absent, 1= occurs sometimes, 2=occurs often) and higher scales indicate greater problems.
Behavior Assessment System for Children (BASC) | pre-intervention, post-intervention (1 week after the completion of the intervention), 3-month follow-up (3 months after the completion of the intervention)
  The BASC is a standardized parent-report of emotional behavior for toddlers and young children.
Brief Observation of Social Communication Change (BOSCC) | pre-intervention, post-intervention (1 week after the completion of the intervention), 3-month follow-up (3 months after the completion of the intervention)
  The BOSCC is a behavioral observation tool originally developed to measure pre- and post-intervention treatment effects in children with autism.
Electroencephalogram (EEG) | pre-intervention, post-intervention (1 week after the completion of the intervention), 3-month follow-up (3 months after the completion of the intervention)
  The Zoo Game will be used as a go/no-go EEG task to measure error-related theta oscillations and error-related negativity (ERN) using EEG tasks.
National Institute for Special Education-Basic Academic Competence Tests (NISE-B ACT) | pre-intervention,post-intervention (1 week after the completion of the intervention), 3-month follow-up (3 months after the completion of the intervention)
  The National Institute for Special Education (NISE) tests will assess basic learning skills, such as reading and math, for students (ages 5 to 14). Higher scores indicate better performance.
Korean-Parent Stress Index-Short Form (K-PSI-SF) | pre-intervention, post-intervention (1 week after the completion of the intervention), 3-month follow-up (3 months after the completion of the intervention)
  The Korean-Parent Stress Index-Short Form is a parent self-report measuring parenting stressors. Higher scores indicate higher levels of parenting stress.

OTHER OUTCOMES:
Barkley Deficits in Executive Functioning Scale (BDEFS) | pre-intervention, post-intervention (1 week after the completion of the intervention), 3-month follow-up (3 months after the completion of the intervention)
  In this study, the Korean version of Barkley Deficits in Executive Functioning Scale (BDEFS) will be used to assess the presence of executive function and attention deficit hyperactivity disorder symptoms in daily lives of caregivers of children with autism.
Kims Frontal Executive Neuropsychology Test (K-FENT) | pre-intervention, post-intervention (1 week after the completion of the intervention), 3-month follow-up (3 months after the completion of the intervention)
  The K-FENT assesses attention, language, visuospatial and memory skills in adults. In this study, the K-FENT will be used to measure EF function of parents.
Emotion Regulation Questionnaire (ERQ) | pre-intervention, post-intervention (1 week after the completion of the intervention), 3-month follow-up (3 months after the completion of the intervention)
  The ERQ will be used to measure how parents experience and express their emotions. Higher scores indicate greater use of that particular emotion regulation strategy.
Loneliness and Social Isolation Scale (LSIS) | pre-intervention, post-intervention (1 week after the completion of the intervention), 3-month follow-up (3 months after the completion of the intervention)
  The LSIS is an instrument that encompasses both objectively measurable "social network" and an individual's subjective perceptions of "social support" and "loneliness" to estimate the complex concept of "social isolation".
UCLA (University of California, Los Angeles) Loneliness Scale | pre-intervention, post-intervention (1 week after the completion of the intervention), 3-month follow-up (3 months after the completion of the intervention)
  The Korean version of the UCLA Loneliness Scale will be used to assess loneliness as 'a state of extreme distress due to relational deficiency'. Higher scores indicate greater levels of loneliness.

CONTACTS AND LOCATIONS:
Overall Officials: So Hyun Kim, PhD, Principal Investigator — Korea University; Boin Choi, PhD, Study Director — Korea University
Locations (1):
- Korea University, Seoul, South Korea